CLINICAL TRIAL: NCT04961281
Title: Dexmedetomidine Versus Triamcinolone Local Injection for Pain Alleviation in Patients With Carpal Tunnel Syndrome; A Randomized Clinical Trial
Brief Title: Dexmedetomidine Versus Triamcinolone Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB0002021
Record Dates: First submitted 2021-06-22; First posted 2021-07-14 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Chronic Pain; Carpal Tunnel Syndrome
MeSH Terms: conditions — Chronic Pain; Carpal Tunnel Syndrome | interventions — Dexmedetomidine; Triamcinolone

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Investigate if, and to what extent,carapl tunnel hydro-dissection using DEX or triamcinolone (TM) along with saline, under ultrasound guidance, can improve the clinical condition, change in nerve conduction parameters of patients with CTS and delay or avoid the surgical intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmeditomidine group (Active Comparator): injection of 1 microgram/kg dexmeditomidine + 10 cc saline injection nearby median nerve as hydro-dissection
  Interventions: Drug: Dexmedetomidine
- triamcinolone group (Active Comparator): injection of 40 mg triamcinolone + 10 cc saline injection nearby median nerve as hydro-dissection
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Dexmedetomidine — injection of Dexmedetomidine ( 10 microgram/kg) + 10 cc saline injection nearby median nerve as hydro-dissection
  Arms: Dexmeditomidine group
Drug: Triamcinolone — injection of triamcinolone ( 40 mg) + 10 cc saline injection nearby median nerve as hydro-dissection
  Arms: triamcinolone group

SUMMARY:
Carpal tunnel syndrome (CTS) is a common mononeuropathy due to entrapment of the median nerve in the carpal tunnel. a lot of modaleties are available for treatment of mild to moderate CTS.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a common mononeuropathy due to entrapment of the median nerve in the carpal tunnel. a lot of modaleties are available for treatment of mild to moderate CTS.

In case of failed conservative oral therapey, local hydro-dessction of the median nerve can be done with saline alone. local anethetics, steroids, hyalase,and ozone have been utilized to augment the symptoms reliefe.

Dexmeditomidine (DEX) has been studied as adjuvant for nerve block to aumnet the pain reliefe. Recently, it has been discovered that DEX can offer some antinflammatory effects when injected in the perineural area. Upon such discovery, the goal of this study has been built.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* complaining of carpal tunnel syndrome of 3 month duration or more
* diagnosed axonal neuropathy using electrodiagnosis , nerve conduction study

Exclusion Criteria:

* patient refusal
* infection at the site of intervention
* allergy to utilized drugs
* diabetic
* previous surgery in the site of injection
* previous injection in the targeted site within the last year

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
pain visual analoge scale | 6 months
  visual analog scale of pain value of (0 cm) no pain , and value of (10 cm) worst pain

SECONDARY OUTCOMES:
change of cross sectional area of the median nerve | 6 months
  change of cross sectional area of the median nerve mm2

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Connor D, Marshall S, Massy-Westropp N. Non-surgical treatment (other than steroid injection) for carpal tunnel syndrome. Cochrane Database Syst Rev. 2003;2003(1):CD003219. doi: 10.1002/14651858.CD003219. PMID 12535461
- [Background] Li B, Li Y, Tian S, Wang H, Wu H, Zhang A, Gao C. Anti-inflammatory Effects of Perioperative Dexmedetomidine Administered as an Adjunct to General Anesthesia: A Meta-analysis. Sci Rep. 2015 Jul 21;5:12342. doi: 10.1038/srep12342. PMID 26196332
- [Background] Brummett CM, Norat MA, Palmisano JM, Lydic R. Perineural administration of dexmedetomidine in combination with bupivacaine enhances sensory and motor blockade in sciatic nerve block without inducing neurotoxicity in rat. Anesthesiology. 2008 Sep;109(3):502-11. doi: 10.1097/ALN.0b013e318182c26b. PMID 18719449
- [Background] Sukegawa S, Higuchi H, Inoue M, Nagatsuka H, Maeda S, Miyawaki T. Locally injected dexmedetomidine inhibits carrageenin-induced inflammatory responses in the injected region. Anesth Analg. 2014 Feb;118(2):473-480. doi: 10.1213/ANE.0000000000000060. PMID 24445644
- [Background] Honda Y, Higuchi H, Matsuoka Y, Yabuki-Kawase A, Ishii-Maruhama M, Tomoyasu Y, Maeda S, Morimatsu H, Miyawaki T. The inhibitory effect of locally injected dexmedetomidine on carrageenan-induced nociception in rats. Eur J Pharmacol. 2015 Oct 5;764:215-219. doi: 10.1016/j.ejphar.2015.06.054. Epub 2015 Jul 6. PMID 26160316